CLINICAL TRIAL: NCT05016713
Title: Changes in Streptococcus Mutans Colonization With Different Oral Hygiene Protocols in Adult Patients With Fixed Orthodontic Appliance:A Randomized Clinical Trial
Brief Title: Changes in Streptococcus Mutans Colonization With Different Oral Hygiene Protocols in Adult Patients With Fixed Orthodontic Appliance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelsalam Ahmed Abdelsalam Elbanna, Master candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 8321
Record Dates: First submitted 2021-08-13; First posted 2021-08-23 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: S.Mutans Colonization in Adults With Fixed Orthodontic Appliance
Keywords: streptococcus mutans; bacterial colonization; fixed appliance; plaque; oral hygiene; orthodontic appliance; adult
MeSH Terms: conditions — Plaque, Amyloid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of the operator: Blinding will not be possible for the operator during the application interventions and during the follow up visits as he will be responsible for recruitment of sample, giving instruction about different hygiene measures that will be used by intervention/control group and follow up of patients collecting samples for that will be used in analysis.
  Blinding of the outcome assessors: It is a single blinded study, the outcome assessors only will be blind. The patients name will be sealed from pre and post samples. Then assessor will carry on, blindly and independently, the measurements and analysis of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention group 1 (Active Comparator): Fluoride-based toothpaste is used for tooth-brushing beside using interdental brushes.
  Interventions: Device: Interdental brush; Other: Fluoride-based toothpaste
- Intervention group 2 (Active Comparator): Chlorhexidine mouthwash is added to the previous oral hygiene protocol being used beside fluoride-based toothpaste and interdental brushes. CHX mouthwash is used by patients according to the manufacturer's instructions 15 min after tooth-brushing: 5 mL of 0.2% CHX was applied for 60s in the morning and at bedtime. The patients will be instructed not to consume any liquid or food at least 30 min after using the prescribed mouthwash. All patients are asked to bring the mouthwash bottle, so we could determine patient compliance based on how much liquid was left.
  Interventions: Combination Product: Chlorhexidine mouthwash; Device: Interdental brush; Other: Fluoride-based toothpaste
- Control group (Placebo Comparator): Regular tooth-brushing is carried out using fluoride-based toothpaste supplied only.
  Interventions: Other: Fluoride-based toothpaste

INTERVENTIONS:
Combination Product: Chlorhexidine mouthwash — Chlorhexidine mouthwash is added to the oral hygiene protocol being used beside fluoride-based toothpaste and interdental brushes. CHX mouthwash is used by patients according to the manufacturer's instructions 15 min after tooth-brushing: 5 mL of 0.2% CHX was applied for 60s in the morning and at bedtime. The patients will be instructed not to consume any liquid or food at least 30 min after using the prescribed mouthwash. All patients are asked to bring the mouthwash bottle, so we could determine patient compliance based on how much liquid was left.
  If any participant shows any signs of CHX hypersensitivity, the intervention will be discontinued.
  Arms: Intervention group 2
Device: Interdental brush — Fluoride-based toothpaste is used for tooth-brushing beside using interdental brushes.
  Arms: Intervention group 1; Intervention group 2
Other: Fluoride-based toothpaste — Regular tooth-brushing is carried out using fluoride-based toothpaste supplied only.

SUMMARY:
Fixed orthodontic appliances increase the rate of plaque accumulation around orthodontic brackets and gingival margins. It was also found that the amount of plaque accumulation and S.mutans level around banded orthodontic appliances is much higher than unbanded appliances.appliances. This increases the importance of regular use of conventional tooth brushing with or without mouthwash for better control of plaque accumulation. Different studies had been conducted to compare the effect of different mouthwashes on plaque accumulation and rate of different bacterial colonization. Among which is Chlorhexidine mouthwash that showed highest antiseptic effect.

S. mutans bacteria are the main reason for the formation of plaque and dental caries associated with the use of fixed braces in 30-70% of patients. It also causes the appearance of white spot lesions on the teeth during and after fixed orthodontic treatment. Therefore, it is necessary to find solutions to overcome the occurrence of these effects resulting from the use of fixed braces, which usually makes it difficult for the accessing of various cleaning tools to these narrow places around the orthodontic brackets. Therefore, it is necessary to find an effective and easy way to clean the teeth that guarantees the safety of the patient's teeth during and after orthodontic treatment.Although mechanical plaque removal is very effective way in controlling amount of plaque accumulation, it is not applicable for subsequent application in patients with fixed orthodontic appliance.

Streptococcus mutans is considered as the main colonizer in the multi-species plaque biofilm. Studies found that as early as one week after bonding of fixed orthodontic appliances, significant changes occurred in the oral microbiota forming microbial plaque at the metal surfaces and the adjacent tooth surface.

The aim of this study is to compare the effect of three different oral hygiene protocols on the amount of Streptococcus mutans colonization in adult patients with fixed orthodontic appliance.

The null hypothesis is that there is no difference on the amount of Streptococcus mutans colonization between using combined tooth brushing, interdental brushing and mouthwash than using tooth brushing and interdental brushing in comparison to tooth brushing alone in adult patients with fixed orthodontic appliance.

DETAILED DESCRIPTION:
The study will take place in the clinic of the Orthodontic Department at the Faculty of Oral and Dental Medicine, Cairo University. The recruited sample will be from the Egyptian population. The principal investigator will recruit the patients according to planned eligibility criteria from the clinic of Orthodontic Department, Faculty of Dentistry, Cairo University. Screening of patients will continue until the total number (27 patients) of participants for the study is collected.

Principal investigator will fill a medical history questionnaire for every patient to exclude the presence of any systemic condition interfering with orthodontic treatment.

Proper examination of the oral structures is needed to identify caries, fracture or missing teeth.

Principal investigator will be carefully examining gingival tissues for any gingivitis, periodontitis, recession or lesions.

Principal investigator will check the potential patient to fulfill the inclusion criteria. Then will ask every participant to sign an informed consent about the study. Full set of records (study models, lateral cephalometric radiographs, photos) will be taken by the principal investigator for every patient as part of the routine procedure for treatment of patients in the outpatient clinic of the Orthodontic Department, Cairo University.

Bonding of upper and lower arches with bracket prescription MBT 0.022-inch (American orthodontics) and bondable tubes on molars.

American Orthodontics O-ties will be standardized for all participants. The orthodontic treatment procedure by implementation of NiTi wires for the alignment and initial leveling stages, followed by stainless steel wires for the subsequent stages.

At the end of the initial bonding appointment, an oral hygiene kit (toothbrush Oral-B soft, fluoride-toothpaste) will be given to all participants. According to BOS oral hygiene leaflet, standardized oral hygiene instructions are given. Participants will be shown how to use the items in the kit followed by participants practicing their use.

In intervention group 1: Fluoride-based toothpaste is used for tooth-brushing beside using interdental brushes.

In intervention group 2: Chlorhexidine mouthwash is added to the previous oral hygiene protocol being used beside fluoride-based toothpaste and interdental brushes. CHX mouthwash is used by patients according to the manufacturer's instructions 15 min after tooth-brushing: 5 mL of 0.2% CHX was applied for 60s in the morning and at bedtime. The patients will be instructed not to consume any liquid or food at least 30 min after using the prescribed mouthwash. All patients are asked to bring the mouthwash bottle, so we could determine patient compliance based on how much liquid was left.

If any participant shows any signs of CHX hypersensitivity, the intervention will be discontinued.

In control group: regular tooth-brushing is carried out using fluoride-based toothpaste supplied only.

According to Silness and Löe (1964) each patient's plaque index (PI) is determined by only the index teeth (tooth numbers: 16, 12, 24, 36,32, and 44). Briefly, determination of PI will be performed as follows: running an explorer along the surfaces of the teeth both supra and subgingivally which give better results than the use of disclosing solution. Prior to examination gingivae and teeth are dried by a blast of air. No cotton is used in order not to interfere with the soft deposits. Each of the four surfaces of the teeth (buccal, lingual, mesial and distal) is given a score from 0-3, score 0 when there is no plaque on the tooth wall, 1 when plaque is invisible to the naked eye but can be collected using a probe, 2 when plaque is visible at the gingival margin, and 3 when plaque not only is visible at the gingival margin but also cover a significant part of the tooth wall. The scores from the four areas of the tooth are added and divided by four in order to give the plaque index for the tooth. The indices for the teeth (incisors, premolars and molars) may be grouped to designate the index for the group of teeth. By adding the indices for the teeth and dividing by six the index for the patient is obtained. The index for the patient is thus an average score of the number of areas examined.

Sample collection: Samples will be taken for both groups at fixed timelines where the quantities of S. mutans will be calculated in the form of colony-forming units (CFU). First sample will be collected immediately before orthodontic brackets bonding (T0). The second sample will be collected four weeks after bonding (T1). Each group of patients will be used to adhering to the prescribed oral hygiene protocol. Participants are asked to refrain from eating and drinking for ≥1 h prior to sample collection, and they are required to rinse their mouths and sit quietly prior to sample collection.

Adherence protocol:

Achieving good communication skills with patients to improve the efficacy of hygiene control strategies is of the utmost importance. For achieving patient adherence to the prescribed oral hygiene protocol prescribed, the patients are motivated by chair-side motivation and active reminder motivation. Chair-side motivation is more formal and professional, focused about unwanted drawbacks of improper oral hygiene to create a sense of being threatened if patients do not follow instructions. Beside intentionally informing the patients that they are enrolled in the study, result in sense of being observed through Hawthorne effect. Moreover, using active reminder motivation allow for patients' compliance to their oral hygiene by a reminder system they prefer. This is achieved by using cell phones to send reminding SMS and app-based text messages to patients or their parents. Setting a WhatsApp-based chatting room for participants to share teeth selfies, this allow for better compliance to oral hygiene through Hawthorne effect.

Data management:

A colleague outside the research team will enter the data and organize it in excel sheets in the computer of the orthodontic department.

Statistical methods:

Results will be sent to a specialized statistician.

The specialized statistician will be responsible for the statistical analysis of the study by:

1. Presenting the data as mean, standard deviation (SD) and Standard error (SE) values.
2. Using Paired t-test to compare between the pre-and post -treatment data for each group then using independent t-test to compare between the groups.

   * For this study, the specialized statistician will use IBM11 SPSS12 Statistics Version 20 for Windows to perform the required statistics.
   * The significance level will be P ≤ 0.05. Highly significant variables are detected when P value is less than 0.01.

Assessors Reliability:

* To achieve high reliability for measurements, the supervisor will choose a well-experienced inter-examiner during the study.
* Each examiner will complete the measurements on a model and will repeat the procedure after one week to assess the intra- and inter-examiner reliability.
* The supervisor will compare the measurements of the two assessors for disagreement with a difference of more than one millimeter.
* The supervisor will evaluate the amount of variation in measurements among and between examiners to test the performance of each assessor.
* The examiner with less reliability will receive additional training but will be replaced during the study.
* The specialized statistician will calibrate the intra and inter-examiner reliability for the measurements of the study by the Intra-class correlation coefficient (ICC). The closer the ICC to 1.0, the higher reliability between assessors. According to Fleiss:" ICC values between 0.7 and 0.9 represent good reliability." The kappa scores between study examiners will be calculated, a range of 0.60-0.80 will represent acceptable reliability.

Data monitoring:

Monitoring of the study will be strictly done by the supervisors periodically. They will monitor all the steps of the followed protocol and find solutions to all troubles that have occurred during the trial performance.

Harms If any harms occur to the patient before entry to the study, it will be reported as unrelated. If it happens after, it will be recorded and documented by the primary investigator. Severity of harms and potential causal relationship with intervention will be addressed.

Audit The trial will be audited by the supervisors in orthodontic department at Cairo university frequently.

Informed consent All the details of the trail and the possibility of recruitment will be clearly introduced to the patients. Each patient signed an informed consent before he or she being recruited into the trial.

Access to data To avoid any disclosure of the resulted data all the members of the research team will have access to the study data besides 2 data investigators will be allowed to access the trial data to be able to investigate our results at any time.

Post-trial care Orthodontic treatment will be continued by the principle investigator until the case is finished or will be referred to other colleague according to orthodontic clinic rules of Faculty of Dentistry, Cairo University.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult patients with age range 18-30 years old.
2. Good to fair oral hygiene indicated by healthy non-inflamed gingiva and absence of carious lesions at the time of recruitment.
3. Full permanent dentition (except third molars).
4. Mild to moderate crowding.
5. Lack of using any mouth rinse for at least 1 month before the initiation of the study, and revealing no sign of sensitivity to mouthwashes.

Exclusion Criteria:

1. Presence of any systemic or infectious diseases.
2. History of antibiotic or hormonal therapy within the past 6 months prior to orthodontic treatment.
3. History of smoking.
4. History of professional cleaning (scaling) within the past 3 days prior to sample collection.
5. Presence of major untreated dental conditions such as untreated carious lesions at baseline.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in amount of Streptococcus mutans colonization | T0: pre-bonding. T1: 1 month after bonding.
  Measure the difference in the amount of Streptococcus mutans colonization in adult patients with fixed orthodontic appliance with/without using chlorohexidine mouthwash. Samples will be collected at fixed timelines pre and during orthodontic treatment.

SECONDARY OUTCOMES:
Change in plaque index score | T0: pre-bonding. T1: 1 month after bonding.
  Measure the difference in plaque index score (0-3) in adult patients with fixed orthodontic appliance with/without using chlorohexidine mouthwash pre and during orthodontic treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of oral & dental medicine Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided